CLINICAL TRIAL: NCT03273868
Title: The Effect of a Single Spinal Manipulation on Cardiovascular Autonomic Activity in Healthy Subjects: a Randomized, Cross-over, Sham-controlled Trial
Brief Title: The Effect of a Single Spinal Manipulation on Cardiovascular Autonomic Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Franco Europeen de Chiropratique (Other)
Collaborators: French chiropractic research fund (Unknown)
Responsible Party: Principal Investigator, Mathieu Picchiottino, Chiropractor, PhD student, Institut Franco Europeen de Chiropratique
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Protocole IFEC 2017-01
Record Dates: First submitted 2017-08-09; First posted 2017-09-06 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Manipulation, Spinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High velocity low amplitude manipulation (Experimental)
  Interventions: Other: High velocity low amplitude manipulation
- Sham manipulation (Sham Comparator)
  Interventions: Other: Sham manipulation

INTERVENTIONS:
Other: High velocity low amplitude manipulation — The researcher manually applies a preload force on the T5/T6 level followed by a single posterior to anterior thrust.
  Arms: High velocity low amplitude manipulation
Other: Sham manipulation — The researcher manually applies a preload force on the right scapula followed by a single lateral thrust.
  Arms: Sham manipulation

SUMMARY:
This study evaluates the effect of a single high-velocity low-amplitude spinal manipulation on both cardiovascular autonomic activity and pressure pain thresholds.

It is a cross-over study, thus each participant will undergo both interventions (spinal manipulation and sham manipulation). Both interventions will be separated by a 48 h wash-out period.

DETAILED DESCRIPTION:
Several systematic reviews have shown that spinal manipulations may have an immediate effect on autonomic nervous system activity (e.g. increase in skin sympathetic nerve activity) and on sensitivity to experimentally-induced pain (e.g. increase in pressure pain threshold).

It is generally unknown i) if these supposed effects last after the immediate post intervention period and ii) if there is a statistical relationship between them, considering that pain and autonomic networks are closely connected and interact at the peripheral, spinal and supra-spinal levels.

The primary aim of the study is to assess every single effect immediatly and at short-term after the intervention.

The secondary aim is to assess the bivariate statistical relationship between cardiovascular autonomic activity and sensitivity to experimentally-induced pain after the intervention.

Cardiovascular autonomic nervous system activity is assessed with both heart rate and systolic blood variabilities

Sensitivity to experimentally-induced pain is measured using pressure pain threshold.

ELIGIBILITY:
Inclusion Criteria:

* First-year chiropractic student at IFEC
* Volunteer
* Healthy (no pain, no disease)

Exclusion Criteria:

* Counter indications to spinal manipulation
* Drugs intakes (pain killers or beta-blockers)
* Food, Caffeine and tobacco intakes during the previous hour
* Alcohol intake and performance of strenuous physical activity the day of the experimentation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Heart rate variability (HRV) | Baseline, + 5 minutes, + 15 minutes, + 30 minutes
  Frequency and Time-domain analyses of HRV from 5-minutes ECG recording
Local (T5) and distal (L4) Pressure pain thresholds (PPT) | Baseline, immediatly after intervention, + 12 minutes, + 25 minutes, + 35 minutes
  The mean of 3 successives PPT in kilopascal

SECONDARY OUTCOMES:
Systolic blood pressure variability | Baseline, + 5 minutes, + 15 minutes, + 30 minutes
  Frequency analysis in the low frequency band of systolic blood pressure variability from 5-minutes recording

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Franco Européen de Chiropraxie, Ivry-sur-Seine, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Picchiottino M, Honore M, Leboeuf-Yde C, Gagey O, Cottin F, Hallman DM. The effect of a single spinal manipulation on cardiovascular autonomic activity and the relationship to pressure pain threshold: a randomized, cross-over, sham-controlled trial. Chiropr Man Therap. 2020 Jan 20;28(1):7. doi: 10.1186/s12998-019-0293-4. eCollection 2020. PMID 31988711